CLINICAL TRIAL: NCT02220699
Title: Screening for Osteoporosis in General Practice. Identifying Patients With Osteoporosis in General Practice by Using the Program Data Capture
Brief Title: Screening for Osteoporosis in General Practice
Status: Completed | Type: Observational
Sponsor: Aalborg University (Other)
Collaborators: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Martin Bach Jensen, GP, Ph.D, Professor at Department of Clinical Medicin, Aalborg University and head of the Research Unit of General Practice in Aalborg, Aalborg University
Other Study IDs: FEA-RN-2014-1
Record Dates: First submitted 2014-08-17; First posted 2014-08-20 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Osteoporosis
Keywords: Ostoporosis; Primary Prevention; Health Promotion; General Practice; Secondary screening; Patients at increased risk of osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
All Danish general practices have a data capture system that collects selected data from the electronic patient record. These data are used for various quality assurance purposes. The aim of the study is to evaluate the quality assurance system/program that identifies patients having an increased risk of osteoporosis.

DETAILED DESCRIPTION:
Background/Method

General practitioners (GPs) have the Sentinel data capture program as an integrated part of their medical record system. The program identifies if a patient has one or more of the following risk factors registered with an ICPC code (International Classification of Primary Care - 2, Wonca International Classification Committee (WICC)):

Alcohol abuse (P15), chronic obstructive pulmonary disease (COPD) (R95), hyperthyroidism (T85), rheumatoid arthritis (L88), fracture (L72, L73, L74, L75 and L76 (age > 50))*, anorexia (P86), glomerulonephritis/ nephropathy (U88), early menopause (ages 40 to 45 and X05), smoker (current/former P17), corticosteroid treatment (at least two prescriptions), body mass index (BMI) (between 10-19).

*L72: radius/ulna fracture, L73: tibia/fibula fracture, L74: hand/foot fracture, L75: femur fracture, L76: NEC (not elsewhere classified) fracture.

The GP can generate a list of his own patients that have an increased risk of osteoporosis with name, personal identification number, age, address, eGFR (estimated glomerular filtration rate), BMI, an indication of which of the above mentioned diagnoses the patient has, and whether the patient had been instructed in calcium and vitamin D intake. In order to generate a list, the GP must have been using ICPC coding for at least 6 months with a minimum of 70% of patient contacts.

The GP can afterwards invite these high-risk individuals for a consultation focussing on osteoporosis prevention.

The Study

The study has initiated in January 2014 including two general practices (Clinic A & B) from the Aalborg Municipality that volunteered to participate. Based on the investigators pilot study the investigators aimed at clinics with approximately 200 patients at risk in each.

Clinic A (www.laegernesloejfen.dk) is located in eastern Aalborg, Denmark. Clinic B (www.lægerneiskalborg.dk) is located in southwest Aalborg, Denmark.

Clinic A and B's lists of patients at an increased risk of osteoporosis is printed and downloaded, along with their ICPC coded diagnoses and data.

The patients' medical records are screened for exclusion criteria. Eligible patients are contacted and asked to come for a consultation regarding the risk of developing osteoporosis. The patients are contacted directly if they visit the clinic anyway; otherwise they are contacted by e-mail or letter.

Patients coming for a consultation are given a questionnaire regarding osteoporosis risk factors in relation to lifestyle, diet, diseases predisposing osteoporosis, fall prophylaxis, and medication. The questionnaire also evaluate the patient's attitude towards being offered preventive examination and treatment by his/hers general practitioner. Patients wanting a consultation, but not wishing to participate in the scientific study are examined and offered treatment equal to the consenting patient according to national standards.

The patients then have a consultation regarding osteoporosis prevention (typically by a nurse). During the consultation the patient's different risk factors are discussed and advice is given regarding fall prophylaxis, diet, calcium and vitamin D. The patient's medication is examined as specified by national guidelines. All patients are then offered referral to a DXA-scan.

Patients that are scanned and classified as having osteoporosis are offered a new consultation regarding osteoporosis treatment and blood tests for secondary osteoporosis screening purposes.

Patients with osteopenia and normal bone mineral density are informed about their test result and if necessary advised to have a new DXA-scan in a few years.

The study is based on the routine identification of patients at risk of osteoporosis found by using the Sentinel data capture program. Intervention is not used in the study, however the patients at risk are offered regular preventive examination according to their risk (DXA-scan). The study analyses data based on the quality assurance work regarding osteoporosis of the general practices.

Patients are informed that participation is completely voluntary and they can withdraw from the study at any time and it will have no bearing on present or future treatment. All participating patients give oral and written informed consent.

Patients not wanting to participate will not be part of the study and only their sex, age, risk factors and reason for exclusion will be registered anonymously in order to evaluate the selection of patients.

Lack of participation in the study will have no consequences on the examination and treatment offered to patients at risk.

ELIGIBILITY:
Inclusion Criteria:

* Patient identified as being at an increased risk of osteoporosis by the data capture system

Exclusion Criteria:

* Known osteoporosis.
* Patients treated with alendronate.
* Patients below 25 years of age.
* Bone metastasis.
* Terminal disease.
* Severe dementia or other disease or condition that is incompatible with participation.
* Bone mineral density scan within the past 3 years.
* Errors in their ICPC coding that leads to the patient being misclassified as having an increased risk of osteoporosis.
* Patients not wanting to participate.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at list at the participating general pracitices who are identified to be at an increased risk of osteoporosis by the data capture program are invited to participate (by direct contact, mail or e-mail)
Sampling Method: Non-Probability Sample
Enrollment: 367 (Actual)
Dates: Start 2014-01; Primary Completion 2014-11 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Number of patients with osteoporosis | 6 weeks after visit at the GP clinic
  Participating patients are referred to a bone mineral density measurement (DXA scan). The exact time depends on the waiting time for bone mineral density Measurements.

SECONDARY OUTCOMES:
Number of patients with osteopenia | 6 weeks after visit at the GP clinic
  At the time of bone mineral density measurement
Cost of identifying a patient with osteoporosis | 2 weeks after bone mineral density measurment
  The total cost from inviting the patients until the patients have finished all examinations, except blood testing for secondary osteoporosis (but not including expenses after treatment for osteoporosis may have begun)

OTHER OUTCOMES:
Patients satisfaction with being contacted to participate in a osteoporosis prevention study | baseline
  Assessed by questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Lægerne Sløjfen (a family medicine clinic), Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No